CLINICAL TRIAL: NCT06293612
Title: Role of Microenvironment Analysis and MRI Radiomic Study in the Risk Stratification of Distant Metastases in Rectal Cancer
Brief Title: Constructing a Multimodal Imaging System to Predict the Risk of Heterochronous Metastasis of Rectal Cancer
Acronym: MIS-MRC
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 22/449-3651; 2022-I2M-C&T-B-077 (Other Grant/Funding Number: CAMS Innovation Fund for Medical Sciences (CIFMS)); 7244398 (Other Grant/Funding Number: Youth program of Beijing Natural Science Foundation); Beijing Hope Run Special Fund (Other Grant/Funding Number: LC2021A12)
Record Dates: First submitted 2024-02-18; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Rectal Cancer; Distant Metastasis
Keywords: locally advanced rectal cancer; distant metastases; tumor stromal ratio; magnetic resonance imaging; artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — colonoscopic biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: The patients were randomized into a training cohort (n ＝ 211) to train the model. The patients' clinicopathological data were reviewed, including age, sex, obesity, serum carcinoembryonic antigen and cancer antigen 19-9 levels, T- and N-stages evaluated by MRI, yp-T and yp-N stages evaluated by histopathology. The MR-T/N stages of the tumors were assessed by radiologists. The tumor region of interest was manually delineated on high-resolution oblique axial T2WI and generated the VOI using ITK-SNAP. Overall, 1229 features were extracted from each VOI. Biopsy specimens from colonoscopy were sectioned into 5 μm slices and stained with H&E. Areas with both stromal and tumor cells presented on all four sides were selected to evaluate tumor stroma ratio using an automated scoring method with the highest proportion of stromal components in all measured areas recorded.
  Interventions: Other: No intervention was administrated to the two cohorts.
- Validation cohort: The patients were randomized into a validation cohort (n ＝91) to verify the model. The patients' clinicopathological data were reviewed, including age, sex, obesity, serum carcinoembryonic antigen and cancer antigen 19-9 levels, T- and N-stages evaluated by MRI, yp-T and yp-N stages evaluated by histopathology. The MR-T/N stages of the tumors were assessed by radiologists. The tumor region of interest was manually delineated on high-resolution oblique axial T2WI and generated the VOI using ITK-SNAP. Overall, 1229 features were extracted from each VOI. Biopsy specimens from colonoscopy were sectioned into 5 μm slices and stained with H&E. Areas with both stromal and tumor cells presented on all four sides were selected to evaluate tumor stroma ratio using an automated scoring method with the highest proportion of stromal components in all measured areas recorded.
  Interventions: Other: No intervention was administrated to the two cohorts.

INTERVENTIONS:
Other: No intervention was administrated to the two cohorts.

SUMMARY:
The goal of this observational study is to construct a multimodal intelligent model to predict the risk of heterochronous metastasis of rectal cancer, which is helpful for individualized diagnosis and treatment and follow-up planning. The main questions it aims to answer are:

* what are the independent risk factors of distant metastasis (DM) in locally advanced rectal cancer (LARC)
* What is the influence weight of the above factors on the heterochronous metastasis of LARC, and how to build a risk-prediction model

This study will not affect or interfere with the routine medical diagnosis and treatment of participants, and will not increase the cost and risk of participants. Participant's information is protected and identified by a unique code.

DETAILED DESCRIPTION:
Data collection process in strict implementation of special management, the full name of quality control. Special personnel are responsible for collecting clinical images and pathological information of patients in the medical record system, and personal identification data will be used to identify and process, in order to protect the privacy of test patients/participants. At the same time, there is a special person responsible for quality control and source data verification. Participants use the project unified number as the unique identification code, personal data and case information by the sample management personnel input and save, the user only see the individual number, no longer show the participants' name and other personal information. Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information was built. Participants' sample information is stored electronically in a dedicated computer that is not used for other purposes and is provided with a password, which is only available to the person (1 person) who manages the sample. Participants' medical records will be kept at the hospital and will be accessible only to researchers; If necessary, members of the bidding organization, ethics committee or government management department may access the personal data of the participants according to the corresponding authority. The results of the study will be published as statistically analyzed data and will not contain any identifiable participant information.

The sponsor is responsible for implementing and maintaining quality assurance and quality control systems with written Standard Operating Procedures (SOPs) to ensure that trials are conducted and data are generated, documented (recorded), and reported in compliance with the protocol, good clinical practices (GCP), and the applicable regulatory requirement(s). The SOPs should cover system setup, installation, and use. The SOPs should describe system validation and functionality testing, data collection and handling, system maintenance, system security measures, change control,data backup, recovery, contingency planning, and decommissioning. The responsibilities of the sponsor, investigator, and other parties with respect to the use of these computerized systems should be clear, and the users should be provided with training in use. Noncompliance with the protocol,SOPs,GCP, and/or applicable regulatory requirement(s) by an investigator/institution, or by member(s) of the sponsor's staff should lead to prompt action by the sponsor to secure compliance.

According to the morbidity of LARC and the risk of distant metastasis, the sample size is 300, and the follow-up interval is at least 3 years.

Plan for missing data: If the proportion of missing data is very large, such as greater than 95%, the investigators can directly remove this field; At 50~95%, the investigators have two processing methods, one is to remove this field directly; another way is to turn the field into an indicator variable; that is the 0-1 variable. If the field is empty, the field is 0; Otherwise the field is 1. Between 5% and 50% : In this scenario, the investigators need to fill in the missing values. In the process of filling, there are two categories: simple filling and algorithm filling. Simple filling includes: 0 filling, mean filling, median filling, mode filling; Algorithm filling methods such as K Nearest Neighbors (KNN) filling, random forest filling and so on.

Statistics Statistical Product and Service Solutions (SPSS, version 26.0) and R software (version 4.0.5) were used for statistical analyses. Receiver operating characteristic (ROC) curve analysis was used to evaluate the optimum cutoff value of tumor stromal ratio (TSR) in discriminating DM risk based on the maximum Youden index. Heat maps showed the distribution of variables between patients with or without DM within 3 years. The independent DMFS risk factors were determined using Kaplan-Meier (K-M) curves and Cox regression analysis sequentially based on the data of the training cohort. Statistical significance was set at P<0.05. Inter-observer variability was assessed using κ statistics for categorical and ranked variables, and ICC for continuous variables.

TSR assessment Biopsy specimens from colonoscopy were sectioned into 5 μm slices and stained with H&E. Areas with both stromal and tumor cells presented on all four sides were selected to evaluate tumor stroma ratio (TSR) using an automated scoring method. The highest proportion of stromal components in all measured areas was recorded as the final TSR value in this study.

Magnetic Resonance analysis Machine-learning method was used to analyze the MR images, which includ image acquisition and reconstruction, image segmentation, feature extraction and qualification, analysis, and model building.

Pretreatment magnetic resonance (MR) examinations were conducted using 3.0 T scanners with an 8-channel phased-array wrap-around surface coil. An intramuscular injection of 10 mg raceanisodamine hydrochloride was administered to minimize bowel movement unless contraindicated. Sequences acquired included T1-weighted imaging (T1WI), T2-weighted imaging (T2WI) with and without fat saturation, and diffusion-weighted imaging (DWI) .

The tumor region of interest (ROI) was manually delineated slice-by-slice on high-resolution oblique axial T2WI (orthogonal to the rectal lumen) by the first radiologist and subsequently confirmed by the second radiologist with more experience on Insight Segmentation and Registration Toolkit-Standford Network Analysis Project (ITK-SNAP), from which the three-dimensional whole tumor volume of interest (VOI) was obtained. Disagreements were resolved through discussions. The radiologists were blinded to the clinicopathological information. Overall, 1229 features were extracted from each VOI, which can be classified into four categories: (1) shape characteristics; (2) first-order statistical characteristics; (3) texture features; and (4) high-order statistical characteristics.

The extracted features' inter- and intraclass correlation coefficients (ICCs) were calculated to assess the reproducibility of the features. Features with <0.75 ICCs were considered non-stable and were eliminated. Pearson's correlation analysis was used to identify redundant features, and for any two features with a coefficient of 0.9, the one with the larger mean absolute coefficient was eliminated. The least absolute shrinkage and selection operator algorithm (LASSO) was applied to select the most significant predictive parameter from the training cohort, and 5-fold cross-validation was used to perform dimensionality reduction. A signature (i.e. Radscore) was calculated using a linear combination of the final selected features weighted by the respective coefficients.

Model built and validation According to the results of Cox regression, a nomogram (Mr) integrating all independent risk factors except TSR, a TSR nomogram (Mt) integrating all independent risk factors except the Radscore, and a combined model (Mrt) incorporating all the independent risk factors were constructed to predict the 3-year DM risk. The discriminative ability of these models was evaluated and compared using ROC curves. Calibration plots were drawn to explore the calibration ability of the three models. Decision curve analysis was performed to explore the clinical benefits by calculating the net benefit of each decision strategy at each threshold probability.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed non-mucinous LARC (T3~T4, or any T with N1~2, M0) without previous treatment;
* No concomitant malignancies or systemic disease;
* Complete standard neoadjuvant chemoradiotherapy (NCRT) and radical surgery in our institute;
* Underwent rectal MRI and colonoscopy within 2 weeks before NCRT.

Exclusion Criteria:

* Fail to meet any of the inclusion criteria;
* Inadequate MR image quality for analysis, or lack of biopsy tissue for TSR assessment;
* Incomplete clinical data or withdraw before last visit.

A total of 578 eligible LARC cases were initially reviewed, 276 of which were excluded according to the exclusion criteria. Finally, 302 patients were enrolled in this study and randomized into a training cohort (n ＝ 211) and validation cohort (n ＝ 91).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive cases of locally advanced rectal adenocarcinoma who were treated with 5-FU or Capecitabine-based concurrent NCRT and total mesorectal excision at our institute between 2015 and 2018 were retrospectively reviewed.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Heterochronous distant metastasis | Through study completion, an average of 3 years
  Defined as cancer recurrence at sites outside the pelvis based on radiological and/or histopathological evidence.

SECONDARY OUTCOMES:
Distant metastasis-free survival | From the date of surgery to the date of the first detection of distant metastasis, death from any cause, assessed up to 3 years.
  Distant metastasis-free survival (DMFS) was calculated from the date of surgery to the date of the first detection of distant metastasis, death from any cause, or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Zhang, MD, Study Director — National Cancer Center, Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China
Locations (1):
- National Cancer Center, National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No